CLINICAL TRIAL: NCT07107347
Title: Assessment of Right Ventricular Function for Diagnosis and Prognosis After Acute Pulmonary Embolism: a Comparison of Speckle Tracking Strain and Conventional Echocardiographic Parameters
Brief Title: Assessment of Right Ventricular Function After Acute Pulmonary Embolism: a Comparison of Speckle Tracking Strain and Conventional Echocardiographic Parameters
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Roshdy Abdul Satar Mohamed, assistant lecturer, Assiut University
Other Study IDs: STE in pulmonary embolism
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Acute Pulmonary Embolism (PE)
Keywords: acute pulmonary embolism (PE); STE; right ventricle strain; speckle tracking strain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Echocardiographic Assessment:

Performed within 24h of PE diagnosis Conventional parameters: TAPSE, RV FAC, RV/LV ratio, tricuspid S', PASP STE parameters: RV free wall longitudinal strain (RVFWS), global longitudinal strain (GLS) if feasible All measurements averaged over 3 cardiac cycles (sinus) or 5 (AF)

Follow-up data:

ICU/hospital LOS Need for vasopressors/mechanical ventilation In-hospital and 30-day mortality

DETAILED DESCRIPTION:
the study targets patient with acute pulmonary embolism confirmed by CTPA, without hemodynamic instability. within the first 24 hours echocardiography will be conducted, assessment of RV function by conventional measures eg, TAPSE, S', FCA and speckle tracking strain echocardiography.

compare the results and its sensitivity in prediction of clinical outcomes, that will be assessed by follow up the patients for one month regarding length of hospital stay, oxygen/ventilatory support, hemodynamics support and 30 day mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years.
2. Confirmed acute PE (via CT pulmonary angiography).(4,6)
3. Echocardiography performed within 24 hours of diagnosis.

Exclusion Criteria:

1. Pre-existing significant RV dysfunction (e.g., due to chronic pulmonary hypertension, cor pulmonale or congenital heart disease).
2. History of coronary artery disease.
3. Impaired LV systolic function, ejection fraction <50%.
4. Moderate to severe valvular heart disease.
5. Prior document of an episode of pulmonary embolism.
6. Poor acoustic window.
7. Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged more than 18 years old with confirmed pulmonary embolism
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Primary (main): Composite of in-hospital mortality, ICU admission >7 days, or need for mechanical circulatory/ventilatory support. | 30 day follow up

SECONDARY OUTCOMES:
Secondary outcome: Each individual component; echocardiographic parameters as predictors. | 30 day follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt